CLINICAL TRIAL: NCT02140671
Title: To Deliver a Pilot Project on Effective Interventions to Ensure: Diagnostic Accuracy, Management of Risk and Control and Self-management for Asthma Patients.
Brief Title: Launching an Asthma Initiative Designed to Improve Asthma Management and Outcomes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: British Lung Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ORO3112
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Asthma
Keywords: asthma management; anti-inflammatory therapy; compliance; hospital admission; educations; self-management; guidelines; exacerbations; diagnostic accuracy; symptom control
MeSH Terms: conditions — Asthma; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Patients with an asthma diagnosis
- Patients where there is diagnostic doubt

SUMMARY:
Following on from a 10 year study conducted in Finland this study is designed to test the validity and sustainability of an enhanced asthma management model for the UK.

DETAILED DESCRIPTION:
The British Lung Foundation (BLF) aims to work with the governments in the four UK nations to launch an asthma initiative designed to improve asthma management and outcomes. The project incorporates key learning from a 10 year programme in Finland designed to improve asthma care and cap healthcare costs for paediatric and adult populations.

The Finland programme focused on accurate diagnosis, training and education of healthcare professionals and patients and early use of anti-inflammatory therapy. The programme successfully improved medication compliance, reduced asthma hospital admissions, reduced asthma-related benefit claims and reduced the overall cost of asthma to the Finnish Government.

To test the validity and sustainability of an enhanced asthma management model for the UK, the BLF proposes to undertake a pilot initiative in England. The pilot will focus on: improving diagnostic accuracy through analysis of GP asthma registers; increasing asthma education among healthcare professionals; assessment of risk and control of patient's asthma; supportive self-management and education of people with asthma.

It is anticipated that the pilot will lead to measureable and significant improvements in asthma management, including:

* Reduced number of severe exacerbations (asthma hospitalisation, A&E attendance and oral steroid rescue)
* Improved diagnostic accuracy (and reduction of diagnostic doubt)
* Improved implementation of recognised asthma guidelines, including appropriate step wise management of patients

The pilot will also aim to increase the proportion of patients on the asthma register with an asthma management plan and a recorded asthma control test therefore supporting higher levels of control, and will promote peer-to-peer health care professional asthma education and knowledge sharing to establish an asthma-training legacy.

The pilot model will be sustainable and reproducible across England and the devolved nations (Scotland, Wales and Northern Ireland). Whilst the core aspects of an agreed national model will be rolled out across the pilot site, it will be tailored and refined through local collaboration (primary care, secondary care and commissioners) to help attain local targets in line with regional differences, needs and priorities.

Results from the pilot will be reported 15 months after project initiation on site (July/August 2014)

ELIGIBILITY:
Inclusion Criteria:

* Motivated and driven local champions in the area
* High rates of hospital admissions (aged 3-65)
* High asthma prevalence
* High percentage of patients who have had an asthma review in the previous 15 months.

Exclusion Criteria:

-

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient questionnaire will be subject to local refinement in line with local needs, targets and priorities but will assess -
  * Asthma Control e.g. ACT, or ACQ or RCP3
  * Lifestyle - i.e. smoking status
  * Comorbidities
  * Patient perceived adherence
  * Side effects
  The practice and patient reports will be used to characterise the patient in terms of risk and control. They will give a complete picture of the patient's asthma and will be used to identify patients for diagnostic assessment, medical management and education. Patients will then be stratified into Group 1 (patients with asthma) or Group 2 (Patients identified for further diagnostic assessment and/or with diagnostic doubt).
Sampling Method: Non-Probability Sample
Enrollment: 33370 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Exacerbations reduction | 1 year
  An exacerbation is defined (in line with the European Respiratory Society/American Thoracic Society guidelines) as: acute oral steroids, out of hours or Accident and Emergency (A&E) attendance for asthma, or hospitalisation for asthma.
  Rationale for selecting exacerbations as the primary outcome:
  * They are the time of greatest risk to patients and greatest resource use
  * Exacerbations are defined by routinely held data, such as drug prescriptions (oral steroids and out of hours and A&E attendance), hence are reliable when captured in primary care
  * Exacerbations reflect current control and future risk; a reduction in exacerbations indicates an improvement in asthmatic inflammation control and improved use of anti-inflammatory therapy

SECONDARY OUTCOMES:
1. Increased assessment of patients with equivocal diagnoses and reduction of diagnostic doubt (also detailed under process outcomes) | 1 year
2. Hospitalisations ¬- number and rate - coded for: • Asthma • Lower respiratory conditions (including asthma), i.e. "asthma-related" events | 1 year
3. Inhaled corticosteroids adherence | 1 year
4. Referral rate of high-risk patients to local specialist | 1 year
5. British Asthma Guideline adherence: appropriate step-wise management of patients | 1 year

OTHER OUTCOMES:
1. Accident and Emergency (A&E) attendance | 1 year
2. Proportion of patients on each asthma register that have a confirmed asthma diagnosis | 1 year
3. Proportion of patients with an asthma management plan | 1 year
4. Proportion of patients with a recorded asthma control test (ACT) and Royal College of Physician three questions (RCP3) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David Price, Principal Investigator — Reasearch in Real Life Ltd

REFERENCES:
- See also: Related Info — http://www.cprd.com/